CLINICAL TRIAL: NCT04055623
Title: Phase 2a Study of the Expansion and Infusion of Autologous T-Regulatory Cells in Amyotrophic Lateral Sclerosis
Brief Title: T-regulatory Cells in ALS
Acronym: Tregs in ALS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: Massachusetts General Hospital (Other); The Center for Clinical and Translational Sciences (CCTS) Clinical Research Unit at The University of Texas Health Science Center at Houston (Other); North East Amyotrophic Lateral Sclerosis Consortium (Network)
Responsible Party: Principal Investigator, Jason R. Thonhoff, Principal Investigator, Houston Methodist Neurological Institute, The Methodist Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00022167
Record Dates: First submitted 2019-08-12; First posted 2019-08-14 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: ALS (Amyotrophic Lateral Sclerosis)
Keywords: Lou Gehrig's Disease
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Interleukin-2

STUDY DESIGN:
Intervention Model Description: Group 1 entered the first 6-months is the double-blind part of the study where participants are randomized to Treg cell infusions and low dose Interleukin-2 (IL-2) injections OR placebo (inactive) infusions and placebo IL-2 injections and then went into the open label second 6-months of ascending Treg infusions and IL-2 injections.
  Group 2 went directly into the open label six month trial of ascending Tregs infusions. Group 2 was added due to the pandemic and limits on travel and funding.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The study drugs for the first 6-months of the study are (1) Treg cell intravenous (IV) infusions or matching placebo / inactive infusion and (2) subcutaneous interleukin-2 (IL-2) injections or matching placebo / inactive injections; followed by 6-months of Treg infusions and IL-2 injections for all participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Intravenous infusion of Treg cells + Interleukin-2 injections (Experimental): For the first six months: T-regulatory cells taken from a participant will be increased in numbers outside the body in a lab and then returned back to the same participant through intravenous (IV) infusions once per month. The participant will also take Interleukin-2 (IL2) injections three times per week.
  Interventions: Biological: Monthly autologous Treg cells infusions + 3 times per week Interleukin-2 injections
- Intravenous infusion w/Placebo + matching placebo injections (Placebo Comparator): For the first six months: Participants will receive matching placebo or inactive intravenous (IV) infusions once per month. The participant will also take a matching inactive placebo injection three times per week.
  Interventions: Other: Monthly placebo infusions + 3 times per week placebo injections
- 2nd 6-months Open Label: Treg Infusions + IL-2 injections (Experimental): For second six months: All participants will receive their own expanded/increased in numbers Treg cells by monthly infusion plus 3 times per week subcutaneous injections of IL-2.
  Interventions: Biological: Monthly autologous Treg cells infusions + 3 times per week Interleukin-2 injections

INTERVENTIONS:
Biological: Monthly autologous Treg cells infusions + 3 times per week Interleukin-2 injections — For the first 6-months of the study: T-regulatory cells taken from a patient, increased in number in a lab, and returned through monthly intravenous (IV) infusions back to same patient + 3 times per week subcutaneous Interleukin-2 injections
  Other Names: Individualized therapy Treg cell infusions + Interleukin-2 (IL-2); Proleukin is brand name for IL-2
  Arms: Intravenous infusion of Treg cells + Interleukin-2 injections
Other: Monthly placebo infusions + 3 times per week placebo injections — For first 6-months of study: monthly placebo infusions + 3 times per week subcutaneous placebo injections
  Other Names: inactive drug
  Arms: Intravenous infusion w/Placebo + matching placebo injections
Biological: Monthly autologous Treg cells infusions + 3 times per week Interleukin-2 injections — For the second 6-months of the study: all participants will receive T-regulatory cells taken from the patient, that have been increased in number in a lab, and returned through monthly intravenous (IV) infusions back to same patient (Treg cell owner) + 3 times per week subcutaneous Interleukin-2 injections.
  Other Names: Individualized therapy Treg cell infusions + Interleukin-2 (IL-2); Proleukin is the brand name for IL-2
  Arms: 2nd 6-months Open Label: Treg Infusions + IL-2 injections

SUMMARY:
This study is a randomized, placebo-controlled, phase 2a trial to study the biological activity, safety, and tolerability of regulatory T Lymphocytes (Tregs) taken and expanded outside of the body and returned back to the same person whose Treg were removed, given back by IV (intravenously) and in combination with low-dose IL-2 in people with Amyotrophic Lateral Sclerosis (ALS).

DETAILED DESCRIPTION:
Based on data collected in a previous study with a small group of patients, evidence was found to show that interfering with the immune system using Treg cells slowed ALS disease progression. It is known that Treg cell numbers and function are reduced in patients with ALS and in some patients with lower Treg cells, they have a more marked rapid progression of their ALS. For this study, there are two sites (in Houston, Texas and Boston, Massachusetts) in which Tregs will be taken from participants, increased or expanded outside the body, and then re-administered back to the participants from which the Tregs came.

This study has two parts and due to the pandemic two groups [Group 1 and Group 2]:

1. The first period is a 6-month, randomized, placebo-controlled part of the study to study the biological activity, safety, and tolerability of the monthly expanded Tregs administered intravenously (IV) OR placebo (saline) administered intravenously plus subcutaneous low-dose Interleukin-2 (IL-2) OR subcutaneous placebo (saline) injections in 12 adults with ALS. IL2 helps regulate the immune system's white blood cells. [Group 1 only.]
2. The second period is a 6-month OPEN-LABEL part of the study (no placebo) in which all participants will receive their own expanded Treg cells administered intravenously in combination with subcutaneous low-dose IL-2 at the following schedule: single dose of Treg cells twice (once per month with three IL2 injections per week); followed by double the dose of Treg cells twice (once per month with three IL2 injections per week); followed by triple the dose of Treg cells twice (one per month with three IL2 injection per week); followed by a 1 month follow-up safety visit after the last triple dose of Tregs with was received and the last set of IL2 injections three times per week injections. [Group 1 and Group 2.]

Groups:

GROUP 1 will go through the double-blind part of the study (receive either Tregs infusions and IL2 injections OR saline infusions and saline injections) for six months and open label part of the study (receive Treg injections and IL2 injections) for six months.

GROUP 2 will receive only the open label (Tregs infusions and IL2 injections) for six months.

This study is studying whether the enhancement of Treg numbers and function will slow disease progression.

In the first study of Tregs, we completed a single-center, open-label phase I study of Tregs from people with ALS. Tregs were increased outside the body and returned back to the individual Treg owners in multiple doses every 2 to 4 weeks. This early study provided evidence in a small group of patients that treatment with autologous Tregs may be effective in slowing ALS progression.

ELIGIBILITY:
Inclusion Criteria:

* ALS meeting El Escorial criteria for possible, probable, lab-supported probable, or definite ALS.
* At least 18 years old.
* Provided informed consent and authorized use of protected health information (PHI) in accordance with national and local patient privacy regulations.
* Capable of complying with all study procedures, including the study drug delivery procedure, in the Investigator's opinion.
* On a stable regimen of riluzole for at least 30 days at the time of screening. If not on riluzole at the time of study entry, willing to refrain from initiation of the agent for the duration of the trial.
* Patients on edaravone willing to refrain from taking edaravone on the same day as they will receive the Tregs infusion for the duration of the trial. If not on edaravone at the time of study entry, willing to refrain from initiation of the agent for the duration of the trial.
* Medical record documentation of a decline in ALSFRS-R total score of at least two points in the 90 days prior to screening or at least four points over the 180 days prior to screening.
* Forced vital capacity (FVC) ≥65% of predicted capacity for age, height, and gender at screening.
* Patient able and willing to undergo leukapheresis.

Exclusion Criteria:

* Presence of any of the following clinical conditions that would interfere with the safe conduct of the study, as determined by the Investigator:

  * Unstable neurological, cardiovascular, cerebrovascular, pulmonary, renal, hepatic, endocrine, or hematologic disease; active malignancy or infectious disease; or other medical illness.
  * Unstable psychiatric illness defined as psychosis (hallucinations or delusions), unstable major depression or substance abuse within 180 days prior to screening.
  * Persistent asthma, prior history of acute systemic reactions involving immunoglobulin E (IgE)-dependent mechanisms, history of angioedema, or history of anaphylactic reactions to any medication.
* Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than 3 times the upper limit of normal (ULN) at screening.
* Serum creatinine greater than 1.8 mg/dL or creatinine clearance less than 40 mL/min at screening.
* History of or positive test result for human immunodeficiency virus (HIV), hepatitis C virus, or hepatitis B virus (i.e., positive for both hepatitis B surface antigen and hepatitis B core antibody) at screening.
* Tracheostomy.
* If female, breastfeeding, known to be pregnant, planning to become pregnant during the study, or unwilling to use effective contraception for the duration of the trial and for 90 days after treatment.
* If male of reproductive capacity, unwilling to use effective contraception for the duration of the trial and for 90 days after treatment.
* Enrollment in any other interventional study.
* Treatment with another investigational drug, biological agent, or device within 30 days or 5 half-lives of screening, whichever is longer. Patient participation in an observational/non-interventional clinical study is to be discussed with the Medical Monitor.
* Prior gene or cell therapy treatments for ALS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-08-07 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Treg suppressive function in the blood from baseline to week 24. | Baseline and week 24.
  Change in Treg suppressive function on the proliferation of T-effector cells, as measured in percentage at baseline compared to week 24.

SECONDARY OUTCOMES:
Change in Treg numbers in the blood from baseline to week 24. | Baseline and week 24
  Change in Treg numbers in the blood at baseline compared to week 24; measured in % of total CD4+ cells.
Tolerability of Treg infusions for 6 months of treatment | Baseline to week 24.
  Defined as the percentage of participants who complete the 6-month RCT.
Tolerability of ascending doses of Tregs for 6 months of treatment | Baseline to week 24.
  Defined as the percentage of participants who complete the ascending doses of Tregs.

CONTACTS AND LOCATIONS:
Overall Officials: Stanley H. Appel, MD, Study Director — The Methodist Hospital Research Institute; Jason R. Thonhoff, MD, PhD, Principal Investigator — The Methodist Hospital Research Institute; James D. Berry, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital Neurological Clinical Research Institute, Boston, Massachusetts
  - Houston Methodist Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be shared with requests directed to the research clinical investigators.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At the end of the study via data management plan for duration of Treg studies.
Access Criteria: Request to PI.

REFERENCES:
- [Background] Sakaguchi S. Naturally arising Foxp3-expressing CD25+CD4+ regulatory T cells in immunological tolerance to self and non-self. Nat Immunol. 2005 Apr;6(4):345-52. doi: 10.1038/ni1178. PMID 15785760
- [Background] Viglietta V, Baecher-Allan C, Weiner HL, Hafler DA. Loss of functional suppression by CD4+CD25+ regulatory T cells in patients with multiple sclerosis. J Exp Med. 2004 Apr 5;199(7):971-9. doi: 10.1084/jem.20031579. PMID 15067033
- [Background] Dejaco C, Duftner C, Grubeck-Loebenstein B, Schirmer M. Imbalance of regulatory T cells in human autoimmune diseases. Immunology. 2006 Mar;117(3):289-300. doi: 10.1111/j.1365-2567.2005.02317.x. PMID 16476048
- [Background] Bluestone JA, Buckner JH, Fitch M, Gitelman SE, Gupta S, Hellerstein MK, Herold KC, Lares A, Lee MR, Li K, Liu W, Long SA, Masiello LM, Nguyen V, Putnam AL, Rieck M, Sayre PH, Tang Q. Type 1 diabetes immunotherapy using polyclonal regulatory T cells. Sci Transl Med. 2015 Nov 25;7(315):315ra189. doi: 10.1126/scitranslmed.aad4134. PMID 26606968
- [Background] Beers DR, Henkel JS, Zhao W, Wang J, Huang A, Wen S, Liao B, Appel SH. Endogenous regulatory T lymphocytes ameliorate amyotrophic lateral sclerosis in mice and correlate with disease progression in patients with amyotrophic lateral sclerosis. Brain. 2011 May;134(Pt 5):1293-314. doi: 10.1093/brain/awr074. PMID 21596768
- [Background] Zhao W, Beers DR, Liao B, Henkel JS, Appel SH. Regulatory T lymphocytes from ALS mice suppress microglia and effector T lymphocytes through different cytokine-mediated mechanisms. Neurobiol Dis. 2012 Dec;48(3):418-28. doi: 10.1016/j.nbd.2012.07.008. Epub 2012 Jul 17. PMID 22820142
- [Background] Henkel JS, Beers DR, Wen S, Rivera AL, Toennis KM, Appel JE, Zhao W, Moore DH, Powell SZ, Appel SH. Regulatory T-lymphocytes mediate amyotrophic lateral sclerosis progression and survival. EMBO Mol Med. 2013 Jan;5(1):64-79. doi: 10.1002/emmm.201201544. Epub 2012 Nov 9. PMID 23143995
- [Background] Beers DR, Zhao W, Wang J, Zhang X, Wen S, Neal D, Thonhoff JR, Alsuliman AS, Shpall EJ, Rezvani K, Appel SH. ALS patients' regulatory T lymphocytes are dysfunctional, and correlate with disease progression rate and severity. JCI Insight. 2017 Mar 9;2(5):e89530. doi: 10.1172/jci.insight.89530. PMID 28289705
- [Background] Alsuliman A, Appel SH, Beers DR, Basar R, Shaim H, Kaur I, Zulovich J, Yvon E, Muftuoglu M, Imahashi N, Kondo K, Liu E, Shpall EJ, Rezvani K. A robust, good manufacturing practice-compliant, clinical-scale procedure to generate regulatory T cells from patients with amyotrophic lateral sclerosis for adoptive cell therapy. Cytotherapy. 2016 Oct;18(10):1312-24. doi: 10.1016/j.jcyt.2016.06.012. Epub 2016 Aug 3. PMID 27497700
- [Result] Thonhoff JR, Beers DR, Zhao W, Pleitez M, Simpson EP, Berry JD, Cudkowicz ME, Appel SH. Expanded autologous regulatory T-lymphocyte infusions in ALS: A phase I, first-in-human study. Neurol Neuroimmunol Neuroinflamm. 2018 May 18;5(4):e465. doi: 10.1212/NXI.0000000000000465. eCollection 2018 Jul. PMID 29845093
- [Derived] Thonhoff JR, Berry JD, Macklin EA, Beers DR, Mendoza PA, Zhao W, Thome AD, Triolo F, Moon JJ, Paganoni S, Cudkowicz M, Appel SH. Combined Regulatory T-Lymphocyte and IL-2 Treatment Is Safe, Tolerable, and Biologically Active for 1 Year in Persons With Amyotrophic Lateral Sclerosis. Neurol Neuroimmunol Neuroinflamm. 2022 Aug 29;9(6):e200019. doi: 10.1212/NXI.0000000000200019. Print 2022 Nov. PMID 36038262